CLINICAL TRIAL: NCT00439361
Title: Phase-I Study of Bortezomib (VELCADE) Plus ICE (Ifosfamide, Carboplatin, Etoposide) for Patients With Relapsed Classical Hodgkin Lymphoma
Brief Title: Velcade Plus ICE for Patients With Relapsed Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0527
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Hodgkin Lymphoma; Lymphoma
Keywords: Hodgkin Lymphoma; HL; Relapsed Classical Hodgkin Lymphoma; Refractory; Lymphoma; Nodular sclerosis; Mixed cellularity; Lymphocyte-rich classical HL; Bortezomib; Velcade; LDP-341; MLN341; PS-341; Carboplatin; Paraplatin; Etoposide; VePesid®; Ifosfamide; Mesna; Mesnex; ICE
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Bortezomib; Carboplatin; Etoposide; Ifosfamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib + ICE (Experimental): Bortezomib + ICE (Ifosfamide, Carboplatin, Etoposide):
  Bortezomib 1.0 mg/m^2 intravenous (IV) over 5 Seconds on Days 1 and 4; + ICE (Ifosfamide 5 Gm/m^2 IV continuous infusion on Day 1, Carboplatin 5 AUC IV over 1 Hour Day 1, Etoposide 100 mg/m^2 IV over 2 Hours Days 1-3) + Mesna 5 mg/m^2 IV continuous infusion Day 1; 2 Gm/m^2 IV continuous infusion over 12 Hours.
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Drug: Mesna

INTERVENTIONS:
Drug: Bortezomib — 1.0 mg/m^2 by Vein Over 5 Seconds on Days 1 and 4
  Other Names: Velcade; LDP-341; MLN341; PS-341
Drug: Carboplatin — 5 AUC by Vein Over 1 Hour On Day 1
  Other Names: Paraplatin®
Drug: Etoposide — 100 mg/m^2 By Vein Over 2 Hours On Days 1-3
  Other Names: VePesid®
Drug: Ifosfamide — 5 Gm/m^2 By Vein Continuous Infusion Over 24 Hours On Day 1
Drug: Mesna — 5 mg/m^2 IV continuous Infusion over 24 Hours On Day 1; 2 Gm/m^2 IV continuous infusion over 12 hours starting after completion of Ifosfamide + Mesna 24 hour continuous infusion
  Other Names: Mesnex

SUMMARY:
Primary Objectives:

1. To determine the toxicity profile of multiple doses of bortezomib when given with ICE in patients with relapsed and refractory classical Hodgkin lymphoma (HL).
2. To determine the maximum tolerated dose (MTD) of bortezomib when given in combination with ICE chemotherapy in patients with relapsed and refractory classical Hodgkin lymphoma (HL).

Secondary Objectives:

- To determine the overall response rate and complete response rate in patients with relapsed and refractory classical Hodgkin lymphoma (HL).

DETAILED DESCRIPTION:
Bortezomib is designed to block a protein that plays a role in cell function and growth, which may cause cancer cells to die.

ICE is a combination of chemotherapy drugs that, together, may work more effectively at causing cancer cells to die by stopping cells from dividing.

Mesna is a drug that protects bladder cells from damage by the chemotherapy drug ifosfamide. It is used to decrease the risk of bleeding in the bladder.

Before you can start taking the drugs on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. These tests may be performed within 28 days of starting the study drugs. If you have had some of these exams, tests, or procedures performed recently, they may not need to be repeated. This will be for your study doctor to decide. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight. You will have x-rays and a bone marrow biopsy to check the status of the disease. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. You will have a computed tomography (CT) scan of your abdomen, chest, and pelvis and a positron emission tomography (PET) scan. Blood (about 2-3 tablespoons) will be drawn for routine tests. Women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test within 1 month before starting therapy on this study. Because taking part in this study requires that participants' ability to fight off infections be normal, you will have blood drawn (about 1-2 tablespoons) to be tested for HIV within 6 months before starting therapy on this study. If your HIV test results are found to be positive, you will not be able to take part in this study.

All participants will receive bortezomib as a fixed dose, which will not change unless any intolerable side effects occur. At the start of this study, 3 participants will be given a dose of bortezomib. If this dose does not cause intolerable side effects, the dose will be increased as new participants take part in this study. There will be a total of 3 groups (with 3-6 participants per group) entered at increasing dose levels. The dose of bortezomib you receive will depend on when you join this study.

If you are found to be eligible to take part in this study, you will receive bortezomib plus ICE by vein. You will receive bortezomib, on Days 1 and 4, over 5 seconds. The ICE regimen will be given as a continuous infusion over different times as follows. On Day 1, you will receive ifosfamide and mesna over 24 hours. On Day 2, you will receive mesna over 12 hours and carboplatin over 1 hour. On Days 1-3, you will receive etoposide over 2 hours. This schedule for bortezomib plus ICE is considered 1 cycle (2 weeks) and will be repeated every 14 days.

You may have 3-6 cycles of the study drugs, depending on your tolerance of the drugs and the status of the disease. If the disease gets worse or you experience any intolerable side effects, you will be taken off this study.

Blood (about 2-3 tablespoons) will be drawn once a week for routine tests. You will have a study visit before the start of each 2-week cycle. During these visits, you will have a brief questionnaire that will ask about specific side effects you might be experiencing. It should take about 5 minutes to complete this questionnaire.

After completing 3 cycles, you will return for CT scans, bone marrow biopsies (if they were positive for disease before you began on this study), and a PET scan to check the status of the disease.

After completing 3 cycles (if the disease did not worsen and intolerable side effects did not occur), you may continue on this study for 3 more cycles. During Cycles 4-6, you will have the same scans and blood tests as mentioned above.

After completing this study, for every 3-4 months on an indefinite basis, you will have follow-up visits. During these visits, you will have blood drawn (about 2-3 tablespoons) for routine tests. You will also have the same scans that were performed during the screening visit.

This is an investigational study. Bortezomib and ICE are FDA approved and commercially available. The combination of bortezomib plus ICE is considered investigational and authorized for use in research only.

Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory classical Hodgkin lymphoma (nodular sclerosis, mixed cellularity, or lymphocyte-rich classical HL).
* Patients must have failed front-line standard anthracycline-containing regimen, such as ABVD, Stanford V, or BEACOPP.
* Bidimensionally measurable disease with at least 1 lesion >/= 2.0 cm in a single dimension
* Acceptable hematologic status: Hemoglobin >/= 8.0 g/dL; Absolute neutrophil count >/= 1500 cells/mm^3; Platelet count >/= 100,000 cells/mm^3
* Pre-study World Health Organization (WHO) performance status of 0, 1, or 2
* Age greater than or equal to 16 years
* Voluntary signed IRB approved consent informed before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patients of reproductive potential must follow accepted birth control methods during treatment and for 3 months after completion of treatment. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study. Female patients must not be pregnant or lactating.

Exclusion Criteria:

* Lymphocyte predominant histology
* More than one prior chemotherapy regimen.
* Prior stem cell transplant
* Abnormal liver function:Bilirubin > 2.0 mg/dL (26 µmol/L); Alkaline phosphatase > 2 * upper limits of normal (ULN); AST (SGOT) > 2 * ULN
* Serum creatinine > 1.5 mg/dL (177 µmol/L) within 14 days before enrollment
* Presence of CNS involvement with Hodgkin lymphoma
* Presence of HIV infection or AIDS
* Patient has >/= Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to boron or mannitol.
* Prior bortezomib therapy.
* Another primary malignancy (other than squamous cell and basal cell carcinoma of the skin, in situ carcinoma of the cervix, or treated prostate cancer with a stable PSA) for which the patient has not been disease-free for at least 3 years
* Serious nonmalignant disease (e.g., congestive heart failure, hydronephrosis); active uncontrolled bacterial, viral, or fungal infections; or other conditions which would compromise protocol objectives in the opinion of the investigator and/or the sponsor.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerable Dose (MTD) of Bortezomib when given in combination with ICE chemotherapy in participants with relapsed and refractory classical Hodgkin lymphoma (HL) | Two-week cycle
  MTD dose escalation stops either at the highest indicated dose of bortezomib (1.5 mg/m2), or when a Dose limiting toxicity (DLT) has been observed in at least one third of the patients at any dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A. Fanale, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org